CLINICAL TRIAL: NCT06276803
Title: The LINFU® U.S. Registry for the Detection of Low and High-Grade Atypia and Early, Asymptomatic Pancreatic Ductal Adenocarcinoma (PDAC) in the General Population Without Risk Factors
Brief Title: The LINFU® U.S. Registry for the in the General Population Without Risk Factors
Status: Not yet recruiting | Type: Observational
Sponsor: Adenocyte, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Adenocyte 104
Record Dates: First submitted 2024-02-18; First posted 2024-02-26 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma; Pancreatic Dysplasia
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Slides and cell blocks made from pancreatic fluid collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who have no risk factors for PDAC: In this study, LINFU® will be evaluated to help identify pancreatic intraepithelial neoplasia-2 (PanIn-2), pancreatic intraepithelial neoplasia-3 (PanIn-3), and early, asymptomatic pancreatic ductal adenocarcinoma (PDAC) in patients with no risk factors and who do not display signs or symptoms of pancreatic disease.
  Interventions: Diagnostic Test: LINFU®

INTERVENTIONS:
Diagnostic Test: LINFU® — Patients will undergo low intensity non-focused ultrasound excitation of the pancreas for a total of 15 minutes using a GE LOGIQ10 or other FDA approved, FDA cleared or FDA exempt ultrasound insonation. A contrast agent will be administered IV during the ultrasound insonation and the patient will also receive a dose of secretin. The pancreatic juice will then be collected for a total of 15 minutes.

SUMMARY:
Adenocyte has developed LINFU®, (Low Intensity Non-Focused Ultrasound excitation of the pancreas) as a method of identifying early, asymptomatic pancreatic cancer and its noninvasive precancerous lesions.. In this study, LINFU® will be evaluated in the general population with no risk factors and who exhibit no signs or symptoms of disease, This study will help determine if LINFU® can be used to help identify early, asymptomatic pancreatic ductal adenocarcinoma (PDAC) or their precursor lesions (PanIn-2, PanIn-3).

DETAILED DESCRIPTION:
Adenocyte has developed a proprietary pancreatic cancer detection method, LINFU®, (Low Intensity Non-Focused Ultrasound excitation of the pancreas) to increase the sensitivity of pancreatic juice cytology. LINFU® consists of analysis of pancreatic fluid collected with the help of low intensity non-focused ultrasound excitation of the pancreas. A contrast agent will be used to create bubbles and possibly increase the number of pancreatic cell we collect for the study. Secretin is also used to increase the number of pancreatic cell excretion to maximize the number of cells collected. A neural network-based computer-assisted system may be used to enhance the analysis of specimens.

In this registry, LINFU® will be studied in patients with no risk factors and who exhibit no signs or symptoms of disease. In this registry, a standardized Case Report Form will be completed for every subject enrolled. Information obtained at baseline will include patient history, clinical and demographic information. The results of all diagnostic tests, surgeries, and biopsies performed after the LINFU® technique for a period of 5 years will be recorded and maintained as clinical registry data. This includes testing and procedures received since enrollment including endoscopic ultrasound-fine-needle aspiration (EUS- FNA),magnetic resonance imaging / magnetic resonance cholangiopancreatography (MRI/MRCP), endoscopic retrograde cholangiopancreatography (ERCP), computed tomography (CT), contrast-enhanced ultrasound (CEUS), treatments performed, pathology results, and pancreatic disease history since enrollment.

The registry case report form is the primary data collection instrument for the registry. All data requested on the form must be recorded and these forms will be monitored carefully by the sponsor to ensure they are completely filled out properly.

ELIGIBILITY:
Inclusion Criteria:

1. Both males and females will be enrolled and must be at least 18 years of age and under age of 90
2. Patients, who in the opinion of the Investigator, do not exhibit any symptoms of PDAC including jaundice, nausea and vomiting, weight loss, abdominal pain, bloating or the feeling of fullness, itchy skin, lower back pain, light-colored, greasy stools, sudden onset type 2 diabetes, etc.
3. Patients, who in the opinion of the Investigator, do not have an abnormal imaging study suggestive of PDAC
4. Patients, who in the opinion of the Investigator, should not be ordinarily screened for PDAC because they do not have risk factors including chronic pancreatitis, family history of PDAC, or genetic cancer syndromes which increase the risk of developing PDAC
5. Institutional Review Board (IRB)-approved consent must be signed by patients to participate in this study.

Exclusion Criteria:

1. Patient under the age of 18 and over the age 90
2. Contraindications to LINFU®/EUS/ERCP as determined by study investigators:

   1. Patient with uncorrectable coagulopathy
   2. Patient that cannot undergo anesthesia due to cardiopulmonary contraindication as deemed by the anesthesiologist
   3. Unstable medically (cardiopulmonary, neurologic, or cardiovascular status)
3. Patients, who in the opinion of the Investigator, are at risk of PDAC because they exhibit any of the following: clinical symptoms of PDAC, imaging abnormalities suggestive of PDAC, genetic syndromes which increase the risk of PDAC, a first degree relative with a history of pancreatic cancer, excessive exposure to dry-cleaning and metalworking chemicals
4. Patients who consume alcohol (greater than 3 drinks/day >1 year or >15g/day for >1 year will be excluded
5. Patient with any history of adult-onset diabetes will be excluded
6. Patients who are obese (body mass index [BMI] of 30 or more) will be excluded
7. Patients who have consumed tobacco in the past for greater than 1 year or current smokers will be excluded.
8. Patients with a history of any pancreatic disease, including chronic pancreatitis, or any pancreatic imaging abnormality including intraductal papillary mucinous neoplasm of the pancreas (IPMN)
9. Patients with baseline lipase levels that are abnormal
10. Pregnant females will be excluded
11. Patient that is unable to provide informed consent
12. Patient with known allergy to the microbubble contrast agent or secretin

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who do not exhibit any symptoms of PDAC, do not have an abnormal imaging study suggestive of PDAC and who do not have risk factors which increase the risk of developing PDAC.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2034-09-15 (Estimated); Study Completion 2034-12-15 (Estimated)

PRIMARY OUTCOMES:
The number of pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified with LINFU® | 5 years
  The total number of asymptomatic pancreatic ductal adenocarcinomas and their noninvasive precursor lesions (PanIn-2, PanIn-3) identified with LINFU® by analysis of pancreatic fluid will be recorded.
The change in size of pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified with LINFU® will be determined long term | 5 years
  Patients with early pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified with LINFU® will be monitored long- term (5 years) by EUS- FNA, MRI/MRCP, ERCP, CT and CEUS to assess whether these tumors increase in size (measured in mm) and to determine how many require medical or surgical intervention.

SECONDARY OUTCOMES:
Determine the number of patients with early pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified with LINFU® that require medical or surgical intervention | 5 years
  Patients with early pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified with LINFU® will be monitored long- term (5 years) by standard imaging studies (EUS- FNA, MRI/MRCP, ERCP, CT and CEUS) to assess whether these tumors increase and to determine how many require medical or surgical intervention.

OTHER OUTCOMES:
Yearly survival rate of patients with early pancreatic ductal adenocarcinomas or their noninvasive precursor lesions identified with LINFU® | 5 years
  Patients will be followed by standard imaging studies (EUS- FNA, MRI/MRCP, ERCP, CT and CEUS) and yearly survival rates of patients with early pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified with LINFU® will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Haber, MD FRCP, Principal Investigator — Manhattan Endoscopy Center

IPD SHARING:
Plan to Share IPD: No